CLINICAL TRIAL: NCT03098862
Title: PREVAIL VI: Identification of Host Genetic Factors Underlying Ebola Virus Disease Risk, Mortality, Long-term Sequelae, Viral RNA Persistence, Humoral Immunity, and Ebola Vaccine Response
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917077; 17-I-N077
Record Dates: First submitted 2017-03-30; First posted 2017-04-04 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Ebola Virus Disease
Keywords: Ebola Virus; Genome-Wide Association Study; Liberia; Ebola Survivors; Ebola Contacts; Natural History
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Direct EBOV exposure risk controls
- 2: EVD fatal cases
- 3: EVD survivor cases
- 4: No known EBOV exposure population controls

SUMMARY:
Background:

Genes are instructions that tell the body how to work and grow. They can affect how the body responds to infection. Researchers want to learn more about genes that affect how the body responds to the Ebola virus. Some people with Ebola get very sick and die. Others do not. The research may lead to better treatments for Ebola virus and other germs.

Objective:

To look for genes that may be related to a person s chance of getting very sick after coming in contact with the Ebola virus.

Eligibility:

People at least 3 years of age who either:

Had Ebola

Had close contact with someone who had Ebola

Were in an Ebola vaccine study

Design:

Participants will have a small amount of blood taken from an arm vein by a needle.

Researchers will collect participants data from other vaccine studies they may have been in.

Participants may be asked questions about their health and social history.

Some participants will have their blood tested for the infection syphilis and HIV, the virus that causes AIDS. Participants will be told the results and will get help finding care, if necessary.

Some participants will have their blood sample tested to see if they have had Ebola in the past.

Blood samples will be stored for future research. They will be marked with a code but not with participants names.

DETAILED DESCRIPTION:
The 2013-2015 Ebola Virus outbreak in Western Africa was unprecedented in size and geographic scope. There were over 28,000 cases and 11,000 deaths. During and following the outbreak, it became evident that spectrum of disease being observed in the communities and the Ebola treatment units was much broader than previously thought. In this study, we aim to identify host genetic factors that underlie the observed variation in disease susceptibility, severity, clinical sequelae, viral persistence, and serological response. We will enroll EVD survivors, close contacts of survivors, EVD healthcare workers, and individuals who have received investigational Ebola vaccines (population controls), and collect a blood sample, HIV/syphilis infection status, demographics, and medical history from participants.

Most subjects will complete study participation after a single study visit; subjects having Ebola serology and/or HIV/syphilis testing done as part of this study will return for one or two follow-up visits to receive their HIV/syphilis test results and post-test counseling and Ebola serology results. We will genotype participants and compare results between cohorts to address the study aims. This may provide insight into pathogenesis and host immunity and potentially suggest new methods of intervention.

ELIGIBILITY:
* INCLUSION CRITERIA:
* EVD Survivor:

  * At least 3 years of age
  * Positive EBOV serology or documented RT-PCR positive status
  * Willing to allow storage of biological samples for future research purposes
* Direct EBOV exposure control:

  * At least 3 years of age
  * Meets at least 1 of the following:

    * Household member, family member, friend, care-provider, or sexual partner of survivor who was in close-contact with the survivor within 3 weeks of the EVD event, and has no history of an ETU stay or treatment for EVD at a CCC or holding center
    * Healthcare worker who participated in treatment of EVD patients with no history of an ETU stay or treatment for EVD at a CCC or holding center
    * Participant in PREVAIL III enrolled as a close-contact
  * Willing to allow storage of biological samples for future research purposes even if he/she withdraws from the study.
* No known EBOV exposure population controls:

  * At least 3 years of age.
  * Meets at least 1 of the following:

    * Enrolled in PREVAIL I
    * Enrolled in PREVAC/PREVAIL V
  * Willing to allow storage of biological samples for future research purposes

EXCLUSION CRITERIA:

* Severe illness from current illness (e.g. malaria) requiring treatment that would be compromised by enrollment in this study. Individuals excluded due to current illness can be enrolled following recovery.
* Any condition in the judgement of the study staff that would make the volunteer unable to participate in the study.
* Incapacity to provide consent, e.g., because of decisional impairment.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EVD survivors, close contacts of survivors, EVD healthcare workers, and individuals who have received investigational Ebola vaccines (population controls)
Sampling Method: Non-Probability Sample
Enrollment: 4830 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Identify genetic variation associated with risk of contracting clinical Ebola Virus Disease when directly exposed to the Ebola virus | At Enrollment
  Disease susceptibility and specific symptoms following EBOV infection
Identify genetic variation associated with mortality from Ebola VirusDisease | At Enrollment
  Disease susceptibility and specific symptoms following EBOV infection

SECONDARY OUTCOMES:
Identify genetic variation associated with post recovery Ebola viral RNA persistence in bodily fluids | At Enrollment
Identify genetic variation associated with the presence of uveitis among EVD survivors identified in PREVAIL III | At Enrollment
Identify genetic variation associated with the magnitude and duration of anti-EBOV IgG titer in both EVD cases and vaccine recipients enrolled in PREVAIL I or PREVAC/PREVAIL V trials | At Enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hensley, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (4):
- Liberia (4):
  - PREVAIL C. H. Rennie Hospital, Kalkata
  - PREVAIL JFK Medical Center, Monrovia
  - PREVAIL Redemption Hospital, Monrovia
  - PREVAIL Duport Road Clinic, Paynesville

REFERENCES:
- [Background] Rasmussen AL, Okumura A, Ferris MT, Green R, Feldmann F, Kelly SM, Scott DP, Safronetz D, Haddock E, LaCasse R, Thomas MJ, Sova P, Carter VS, Weiss JM, Miller DR, Shaw GD, Korth MJ, Heise MT, Baric RS, de Villena FP, Feldmann H, Katze MG. Host genetic diversity enables Ebola hemorrhagic fever pathogenesis and resistance. Science. 2014 Nov 21;346(6212):987-91. doi: 10.1126/science.1259595. Epub 2014 Oct 30. PMID 25359852
- [Background] Leroy EM, Baize S, Volchkov VE, Fisher-Hoch SP, Georges-Courbot MC, Lansoud-Soukate J, Capron M, Debre P, McCormick JB, Georges AJ. Human asymptomatic Ebola infection and strong inflammatory response. Lancet. 2000 Jun 24;355(9222):2210-5. doi: 10.1016/s0140-6736(00)02405-3. PMID 10881895
- [Background] Baize S, Leroy EM, Georges-Courbot MC, Capron M, Lansoud-Soukate J, Debre P, Fisher-Hoch SP, McCormick JB, Georges AJ. Defective humoral responses and extensive intravascular apoptosis are associated with fatal outcome in Ebola virus-infected patients. Nat Med. 1999 Apr;5(4):423-6. doi: 10.1038/7422. PMID 10202932